CLINICAL TRIAL: NCT00920751
Title: Comparison of on Demand Sedation With Study Method Versus on Demand Sedation With Conventional Method for Performing Colonoscopy for Colorectal Cancer Screening and Surveillance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: East Bay Institute for Research and Education (Other)
Responsible Party: Joseph Leung, MD, Sacramento VA Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: EBIRE-GI-003
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Colorectal Cancer Screening
Keywords: water infusion; air insufflation; colonoscopy; colorectal cancer screening

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Water infusion (Experimental): Water infusion in lieu of air insufflation during colonoscope insertion
  Interventions: Procedure: Water infusion
- Air insufflation (Active Comparator): Conventional air insufflation colonoscopy
  Interventions: Procedure: Air insufflation

INTERVENTIONS:
Procedure: Water infusion — Water infusion in lieu of air insufflation during colonoscope insertion
  Arms: Water infusion
Procedure: Air insufflation — Conventional air insufflation colonoscopy
  Arms: Air insufflation

SUMMARY:
Hypothesis

1. Study method achieves lower requirement for medications
2. Study method increases overall cecal intubation with comparable assessment of current experience and patient willingness to repeat future colonoscopy compared with conventional colonoscopy
3. Study method results in reduction in medication-related (cardiorespiratory) complications, faster turn around of patients, compared with conventional colonoscopy
4. Study method improves bowel preparation and increases polyp pickup rate

Colorectal cancer (CRC) screening for the high and the low risk healthy asymptomatic VA patients is being promoted (VHA directive). Compliance with this Directive will result in an increased number of VA patients undergoing colonoscopy. The demand for colonoscopy far exceeds the capacity available to perform the procedure in the VA system. The conventional practice for colonoscopy at VA facilities across the country is to perform colonoscopy under conscious sedation with air insufflation. Efficiency is governed by the fact that sedated patients require time and space for recovery and these are major limiting factors in the current setting for the use of colonoscopy for CRC screening.

Methods that maintain a high success rate and good patient assessment improve overall compliance for surveillance colonoscopy. Our preliminary experience showed that patients are able to complete successful colonoscopy without sedation in 52% of cases when colonoscopy was aided by a water infusion in lieu of air insufflation method. In this group of patients, the shortened recovery time means a quick turn around of patient and a more efficient endoscopy service. Patients are able to communicate better with the staff and physician regarding their problem and discharge instructions, and not subjected to the amnesic effect of sedation. Next day follow-up of patient by telephone contact which requires commitment of staff time can be obviated.

If this randomized study confirms the success of our preliminary findings and this technique is adopted by more endoscopists, a larger number of VA patients may benefit from less sedation complications and at the same time allow for more efficient colonoscopy screening services.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 50 years old), male and female patients
* Scheduled and consented for screening or surveillance colonoscopy
* Accept randomization to the study or the conventional method
* Agree to complete study questionnaires will be considered for enrollment
* Normal healthy patients or patients with mild systemic disease, ASA 1 or ASA 2

Exclusion Criteria:

* Patients who decline to participate, are unable to give informed consent or to complete the questionnaires due to language or other difficulties will be excluded. Excluded patients will be managed by usual procedures at the Sacramento VAMC

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-03

PRIMARY OUTCOMES:
Primary outcome - success of cecal intubation without sedation | 1 year

SECONDARY OUTCOMES:
Diagnostic yield, patients' current experience, willingness to repeat future colonoscopy, turn around time, and staff rating of satisfaction, and medication-related complications. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sacramento VA Medical Center, Mather, California, United States

REFERENCES:
- [Derived] Leung J, Mann S, Siao-Salera R, Ransibrahmanakul K, Lim B, Canete W, Samson L, Gutierrez R, Leung FW. A randomized, controlled trial to confirm the beneficial effects of the water method on U.S. veterans undergoing colonoscopy with the option of on-demand sedation. Gastrointest Endosc. 2011 Jan;73(1):103-10. doi: 10.1016/j.gie.2010.09.020. PMID 21184876